CLINICAL TRIAL: NCT03981419
Title: A Randomized, Placebo-Controlled, Double-Blind Pilot Study to Evaluate the Effect of GRF6021 on Intracellular Signaling Cascades in Blood Leukocytes and Postoperative Recovery Following Primary Hip or Knee Arthroplasty
Brief Title: A Study to Evaluate the Effect of GRF6021 on Postoperative Recovery Following Primary Hip or Knee Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alkahest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AKST6021-211
Record Dates: First submitted 2019-05-09; First posted 2019-06-10 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Recovery
Keywords: Total hip replacement; Total knee replacement

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GRF6021 (Experimental): Participants received 4 doses of GRF6021, 250 milliliters (mL), intravenous (IV) infusion. The first dose was administered on day before surgery, the next two doses on the day of surgery i.e., within 4 hours before start of surgery (first incision), and then upon arrival in the postoperative care unit (within 5 hours after the first incision) and the last dose was administered on the day after the surgery.
  Interventions: Biological: GRF6021
- Placebo (Placebo Comparator): Participants received 4 doses of GRF6021 matching placebo, 250 mL, IV infusion. The first dose was administered on day before surgery, the next two doses on the day of surgery i.e., within 4 hours before start of surgery (first incision), and then upon arrival in the postoperative care unit (within 5 hours after the first incision) and the last dose was administered on the day after the surgery.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: GRF6021 — for IV infusion
  Arms: GRF6021
Other: Placebo — for IV infusion
  Arms: Placebo

SUMMARY:
This study will evaluate the safety, tolerability and effect of GRF6021 on clinical recovery parameters in participants undergoing primary hip or knee arthroplasty.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind pilot study to investigate the effects of GRF6021, a 5% human plasma protein fraction administered by intravenous (IV) infusion, on intracellular signaling cascades in blood leukocytes in participants undergoing primary hip or knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 50-85 years of age scheduled to undergo primary total hip or knee replacement surgery.
* Estimated glomerular filtration rate ≥ 45 mL/min/1.73 m2 .

Exclusion Criteria:

* Blood coagulation disorders.
* Participants who started chronic anticoagulant therapy (warfarin, heparin, low-molecular weight heparin, or Factor Xa inhibitors) in the last 6 months
* Hypercoagulable state.
* Prior hypersensitivity to any human blood product including plasma.
* Treatment with any human blood product, including transfusions and IV immunoglobulin, during the 6 months prior to screening.
* History of immunoglobulin A or haptoglobin deficiency.
* Major surgery, trauma or injury in the last 3 months or minor surgery in the last 1 month.
* Heart disease or congestive heart failure in the 6 months prior to dosing.
* Poorly controlled hypertension.
* Severe anemia.
* Functional impairment of major joint or lower extremity other than joint undergoing surgery.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2021-01-23 (Actual); Study Completion 2021-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alkahest Medical Monitor, Study Director — Alkahest, Inc.
Locations (1):
- Stanford University Medical Center, Palo Alto, California, United States

REFERENCES:
- [Derived] Gaudilliere B, Xue L, Tsai AS, Gao X, McAllister TN, Tingle M, Porras G, Feinstein I, Feyaerts D, Verdonk F, Sabayev M, Hedou J, Ganio EA, Berson E, Becker M, Espinosa C, Kim Y, Lehallier B, Rawner E, Feng C, Amanatullah DF, Huddleston JI, Goodman SB, Aghaeepour N, Angst MS. Infusion of young donor plasma components in older patients modifies the immune and inflammatory response to surgical tissue injury: a randomized clinical trial. J Transl Med. 2025 Feb 14;23(1):183. doi: 10.1186/s12967-025-06215-w. PMID 39953524

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at one investigative site in the United States from 12 July 2019 to 04 March 2021.
Pre-assignment Details: Participants who were scheduled to undergo primary total hip arthroplasty (THA) or total knee arthroplasty (TKA) were randomized in 1:1 ratio to receive GRF6021 or placebo. A total of 55 participants were screened, out of which 38 participants were enrolled in the study.
Period: Overall Study
Arm/Group | GRF6021 | Placebo
Started | 18 | 20
Intent-to-Treat (ITT) Population (ITT population included all randomized participants.) | 18 | 20
Safety Population (Safety population included all participants who received at least 1 dose of the study treatment.) | 18 | 20
Evaluable Population (Evaluable population included all participants who received all 4 doses of study treatment and in whom all blood samples were collected.) | 18 | 19
Completed | 18 | 19
Not Completed | 0 | 1
Not completed — Due to Coronavirus Disease-2019 (COVID-19) | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT population included all participants who met the inclusion criteria and did not meet the exclusion criteria and were randomized in the study.
Groups:
- GRF6021: Participants received 4 doses of GRF6021, 250 mL, IV infusion. The first dose was administered on day before surgery, the next two doses on the day of surgery i.e., within 4 hours before start of surgery (first incision), and then upon arrival in the postoperative care unit (within 5 hours after the first incision) and the last dose was administered on the day after the surgery.
- Total: Total of all reporting groups
Arm/Group | GRF6021 | Placebo | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.70 (5.86) | 65.40 (8.39) | 67.89 (7.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 17 | 20 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black or African American | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  White | 8 | 16 | 24
  Not Reported | 3 | 1 | 4
  Other | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Effect of GRF6021 on Immune Responses to Surgery as Determined by Cytometry by Time of Flight (CyTOF) on Day 2
Description: CyTOF=multiplexed, high-content immune profiling technology, providing high-resolution surveillance of circulating immune cells & response to GRF6021 infusions on surgical recovery. Blood samples were collected for CyTOF analysis & were stimulated with a series of extracellular ligands to analyze evoked intracellular signaling responses. High-dimensional data results were obtained from CytOF, and analyzed using the immunological elastic net (iEN) algorithm, a penalized regression method particularly adapted for the analysis of highly correlated data, as it eliminates redundant parameters while retaining interrelated parameters. Raw data obtained from each sample was entered into the classification model (iEN algorithm) that generated prediction values (presented below) showing the effect of study treatment on immune response post-surgery. A prediction value of 0 & 1 indicated perfect results (i.e., positive response to treatment) for the placebo & GRF6021 arms, respectively.
Time Frame: Day 2 (before start of surgery and post surgery)
Population: Evaluable population included all participants who received all 4 doses of study treatment and in whom all blood samples were collected. Overall number of participants analyzed is the number of participants available for analysis.
Measure: Median (Inter-Quartile Range); unit: predicted value
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 18
predicted value
  Day 2 (Before Surgery Start) | 0.5692 [0.4559 to 0.6269] | 0.4521 [0.3935 to 0.5975]
  Day 2 (Post Surgery) | 0.5326 [0.5180 to 0.5510] | 0.4471 [0.4310 to 0.4853]

2. Secondary Outcome: Change in Functional Status Using the ActiGraph Wearable Device Providing Measurements for Physical Activity/Function and Sleep
Description: At screening, participants were provided with an ActiGraph wearable device & approximately -7 to -3 days before surgery, they were instructed to wear the device. ActiGraph wearable device was used to monitor participants' physical activity, mobility & sleep. Functional status including heart rate & sleep time were collected during the study period except perioperative times when it was removed for surgery. ActiGraph high-dimensional data was analyzed using a standard EN algorithm which utilizes a penalized regression method particularly adapted to the analysis of highly correlated data, as it eliminates redundant parameters while retaining interrelated parameters. Raw data obtained over the entire observation period was entered into a classification model (iEN algorithm) that generated prediction values (presented below) for functional status changes. A prediction value of 1 &2 indicated perfect results (i.e., positive response to treatment) for GRF6021 & placebo groups, respectively.
Time Frame: Baseline; Day 1, Day 3 up to approximately Day 46
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: predicted value
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 18
predicted value | 1.7007 [1.6314 to 1.7200] | 1.3861 [1.3289 to 1.5009]

3. Secondary Outcome: Effects of GRF6021 on Plasma Proteomics
Description: Blood samples collected were analyzed using the Somalogic SomaScan platform which provides a broad overview of proteomics changes by measuring approximately 7,000 proteins. It uses a highly multiplexed and high throughput aptamer-based proteomic technology and deoxyribonucleic acid (DNA)-microarray-based detection. It provides concentration domain values as relative fluorescence units (RFUs). Proteomics high-dimensional data was analyzed using a standard EN algorithm which utilizes a penalized regression method particularly adapted to the analysis of highly correlated data, as it eliminates redundant parameters while retaining interrelated parameters. Raw data obtained from each sample was entered into a classification model (iEN algorithm) that generated prediction values for proteomics which are presented in the data table. A prediction value of 1 and 2 indicated perfect results (i.e., positive response to treatment) for the GRF6021 and the placebo group, respectively.
Time Frame: Pre-infusion on Day 1 (baseline), 2 (before start of surgery and post surgery), and Day 3
Population: as for outcome 1
Measure: Mean (Inter-Quartile Range); unit: predicted value
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 18
predicted value
  Day 1 (Baseline) | 1.4320 [1.2641 to 1.6601] | 1.3716 [1.2417 to 1.7486]
  Day 2 (Before Surgery Start) | 1.4189 [1.2135 to 1.7029] | 1.5245 [1.3442 to 1.6457]
  Day 2 (Post Surgery) | 1.1563 [1.0322 to 1.4885] | 1.7264 [1.4567 to 1.9209]
  Day 3 | 1.3971 [1.1933 to 1.5818] | 1.6284 [1.4737 to 1.9543]

4. Secondary Outcome: Number of Participants With Change From Baseline in Delirium as Assessed Using 3-Minute Diagnostic Interview for Confusion Assessment Method (3-Minute Diagnostic Interview for Confusion [3D-CAM])
Description: The 3D-CAM is a brief verbal assessment tool used to test participants for delirium. Each item in the instrument directly informs one of the 4 CAM features including acute onset of mental status change or fluctuating course of cognition, inattention, disorganized thinking, and altered level of consciousness. For all items on the assessment, the participants answered as "incorrect," "correct," "no," or "yes". The CAM algorithm is considered positive if the following features are present: Feature 1) Acute onset or fluctuating course and Feature 2) Inattention and either Feature 3) Disorganized thinking or Feature 4) Altered level of consciousness. Number of participants at baseline and postbaseline with delirium "present" or "not present" are reported here. The baseline was defined as Day 1 pre-infusion measurement.
Time Frame: Baseline (Day 1 pre-infusion); Days 2 (post-infusion), and 3 (pre-infusion)
Population: Evaluable population included all participants who received all 4 doses of study treatment and in whom all blood samples were collected.
Measure: Count of Participants; unit: Participants
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 19
Participants
  Baseline: Delirium Present | 0 | 0
  Baseline: Delirium Not Present | 18 | 19
  Change from Baseline at Day 2: Delirium Present | 2 | 0
  Change from Baseline at Day 2: Delirium Not Present | 16 | 19
  Change from Baseline at Day 3: Delirium Present | 0 | 0
  Change from Baseline at Day 3: Delirium Not Present | 18 | 19

5. Secondary Outcome: Time to 50% Recovery of Baseline Value on the Surgery Recovery Scale (SRS)
Description: SRS is sensitive & simple tool for assessment of functional recovery following major surgery & consist of 13 items. Impacts on daily activities are scored from 1 (not at all) to 5/6 (all the time). First 8 items were scored from 1 to 6. Rest were scored from 1 to 5. SRS scores were obtained by reversing responses (e.g., 1=6, 2=5, 3=4, 4=3, 5=2 and 6=1) to 5 negatively stated items (items 2, 4, 5, 6, and 7) & then summing across all scale items for an individual at baseline & each scheduled post-baseline time point. SRS total score range=13-63 where higher score indicated better recovery. For postoperative visits 'not applicable' responses were coded into same category as affirmations of 'not at all'. For all other time points 'not applicable' responses were coded as missing data. KM estimate of survival was to be used to summarize time (in Days) from date of randomization to 50% recovery of baseline value in SRS by treatment group. Baseline = Day -7 to -3 pre-infusion measurement.
Time Frame: Baseline; Days 1 and 3 (pre-infusion) and thereafter up to the end of the study (approximately Day 46)
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 19
days | 11.5 [8.0 to 15.0] | 15.0 [8.0 to 24.0]

6. Secondary Outcome: End of Study (EOS) Treatment Comparison of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Description: WOMAC is a widely utilized self-report measure of lower extremity symptoms and function. The WOMAC Likert Scale version used an 11-point scale anchored by the wording "no pain" and "extreme pain" for pain, and "no difficulty" and "extreme difficulty" for physical function. There were 5 questions for pain and 17 questions for physical function (total 22 questions). Scores (maximum 10) for each question of WOMAC were summed for an individual at the End of Study. The calculated scores were used to summarize the WOMAC score by treatment group. For this outcome measure, a full WOMAC score 0-220 point scale was used for data analysis. Higher scores on the WOMAC indicate worse pain and physical functional limitations.
Time Frame: At end of study (approximately Day 46)
Population: Evaluable population included all participants who received all 4 doses of study treatment and in whom all blood samples were collected. Overall number analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 17 | 19
score on a scale | 28.50 (27.39) | 37.30 (38.80)

7. Secondary Outcome: Time to a Score of < 12/40 on a Subset of Questions From the WOMAC, Pain Subscale
Description: WOMAC is a widely utilized self-report measure of lower extremity symptoms and function. The WOMAC Likert Scale version uses an 11-point scale anchored by the wording "no pain" (score=0) and "extreme pain" (score=10) for the pain subscale. The pain subscale consists of 4 items. The total score ranges from 0 (best) to 40 (worse). Higher scores on the WOMAC indicate worse pain. Kaplan Meier (KM) estimate of survival was used to summarize the time (in Days) from the date of randomization to the day when the participant had a non-missing score of < 12. Right-censoring was used to produce Kaplan-Meier time-to-event estimates.
Time Frame: Days 1 and 3 (pre-infusion) and thereafter up to Day 39
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 19
days | 13.5 [8.0 to 22.0] | 16.0 [5.0 to 29.0]

8. Secondary Outcome: Time to a Score of < 18/60 on a Subset of Questions From the WOMAC, Physical Function Subscale
Description: WOMAC is a widely utilized self-report measures of lower extremity symptoms and function. WOMAC Likert Scale version uses an 11-point scale anchored by the wording "no difficulty" (score=0) and "extreme difficulty" (score=10) for physical function subscale. The physical function subscale consists of 6 items. The total score ranges from 0 (best) to 60 (worse). Higher scores on the WOMAC indicate more functional limitations. Kaplan Meier (KM) estimate of survival was used to summarize the time (in Days) from the date of randomization to the day when participant had a non-missing score of < 18. Right-censoring was used to produce Kaplan-Meier time-to-event estimates.
Time Frame: Days 1 and 3 (pre-infusion) and thereafter up to Day 39
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 19
days | 18.0 [11.0 to 22.0] | 18.0 [11.0 to 36.0]

9. Secondary Outcome: Change From Baseline in Mental Health Score in the Short Form-36 (SF-36)
Description: The SF-36 determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 5-8 primarily contribute to the mental component summary (MCS) score of the SF-36. The MCS ranges from 0 (worst) to 100 (best), and higher score indicates better mental health status. Positive change from baseline indicates improvement. The baseline was defined as Day -7 to -3 prior to surgery.
Time Frame: At Baseline and end of study (approximately Day 46)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 19
score on a scale
  Baseline | 56.7 (10.16) | 57.6 (8.50)
  Change From Baseline at End of Study | 2.1 (7.13) | 0.8 (8.62)

10. Secondary Outcome: Change From Baseline in Physical Health Score in the SF-36
Description: The SF-36 determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the Physical Component Summary (PCS) score of the SF-36. The PCS ranges from 0 (worst) to 100 (best), and a higher score indicates better physical condition. Positive change from baseline indicates improvement. The baseline was defined as Day -7 to -3 prior to surgery.
Time Frame: At Baseline and end of study (approximately Day 46)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 19
score on a scale
  Baseline | 32.7 (6.87) | 34.9 (9.68)
  Change From Baseline at End of Study | 4.0 (7.92) | 3.3 (9.90)

11. Secondary Outcome: Change From Baseline in the Beck Depression Inventory-II (BDI-II)
Description: The BDI-II is a 21-item questionnaire used to assess depression. Most items are rated on a 4-point scale from 0 to 3, and a few items are rated on a 7-point scale. Individual item scores are added to get a total BDI-II score from 0 to 63. The higher the total score, the more severe the depression, and the lower the total score, the less severe the depression. A negative change from baseline indicated an improvement. The baseline was defined as Day -7 to -3 prior to surgery.
Time Frame: At Baseline and end of study (approximately Day 46)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 18
score on a scale
  Baseline | 7.3 (9.47) | 5.1 (5.47)
  Change From Baseline at End of Study | -3.2 (9.28) | -2.7 (5.65)

12. Secondary Outcome: Number of Participants With Opioid Analgesic Consumption During Hospital Stay and After Discharge to End of Study
Time Frame: From Day 2 (post-surgery) up to end of study (approximately Day 46)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 19
Participants | 18 | 19

13. Secondary Outcome: Time to Discharge
Description: The Kaplan-Meier (KM) estimate of survival was used to summarize the time (in Days) from the date of randomization to discharge from the hospital by treatment group using median and inter quartile ranges: Q1 (25th percentile) and Q3 (75th percentile).
Time Frame: Day 1 up to end of study (approximately Day 46)
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 19
days | 2.0 [2.0 to 2.0] | 2.0 [2.0 to 2.0]

14. Secondary Outcome: Perioperative Outcome: Surgery Duration
Description: The duration (in hours) for which a participant underwent surgery i.e., primary hip or knee arthroplasty is reported here.
Time Frame: Day 2
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 19
hours | 1.8 [1.1 to 2.4] | 1.6 [1.3 to 2.1]

15. Secondary Outcome: Perioperative Outcome: Duration for Which Participants Were Under Anesthesia
Description: The duration (in hours) for which a participant was under anesthesia is reported here.
Time Frame: Day 2
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 19
hours | 3.0 [2.3 to 4.6] | 2.7 [2.3 to 4.6]

16. Secondary Outcome: Perioperative Outcome: Duration of Stay in the Post-Anesthesia Care Unit (PACU)
Description: The duration (in hours) for which the participants stayed at the PACU is reported here.
Time Frame: Day 2
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 19
hours | 2.6 [1.6 to 5.3] | 2.9 [1.5 to 8]

17. Secondary Outcome: Perioperative Outcome: Number of Participants in Each 5 American Society of Anesthesiologists (ASA) Class
Description: ASA class ranges from ASA I - ASA VI. Higher ASA class with other factors (surgery type, frailty, and deconditioning) help predict greater perioperative risk. Normal healthy participants are categorized under ASA I, whereas participants with mild systematic disease and severe systematic disease are graded as ASA II and ASA III, respectively. If participants have severe systematic disease that is a constant threat to their life, they are graded as ASA IV. A moribund participant who is not expected to survive without the operation is classified as ASA V. ASA VI includes participants that are declared brain-dead and whose organs are being removed for donor purposes.
Time Frame: Day 2
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 19
Participants
  ASA I | 0 | 0
  ASA Il | 8 | 12
  ASA III | 10 | 7
  ASA IV | 0 | 0
  ASA V | 0 | 0

18. Secondary Outcome: Perioperative Outcome: Estimated Blood Loss
Time Frame: Day 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 19
mL | 113.6 (60.00) | 135.8 (96.63)

19. Secondary Outcome: Number of Participants in Whom Intraoperative Fluids Were Administered
Description: Intraoperative fluids administered were summarized by WHO Drug Dictionary (WHO-DD) Version 2018 Anatomical Therapeutic Chemical (ATC) level 3 terms and standardized medication names.
Time Frame: Day 2
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 19
Participants | 0 | 0

20. Secondary Outcome: Number of Participants in Whom Intraoperative Blood Products Were Administered
Description: Intraoperative blood products administered were summarized by WHO-DD Version 2018 ATC level 3 terms and standardized medication names.
Time Frame: Day 2
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 19
Participants | 0 | 0

21. Secondary Outcome: Number of Participants Who Received Intraoperative Anesthesia
Description: Intraoperative anesthesia administered were summarized using WHO-DD Version 2018 ATC level 3 terms and standardized medication names.
Time Frame: Day 2
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 19
Participants
  General Anesthesia | 18 | 19
  Local Anesthesia | 15 | 19

22. Secondary Outcome: Number of Participants Who Received Intraoperative Opioids
Description: The number of participants with intraoperative opioids administered were summarized by WHO-DD Version 2018 ATC level 3 terms and standardized medication names.
Time Frame: Day 2
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 19
Participants
  Oxycodone | 17 | 19
  Hydromorphone | 9 | 6
  Hydrocodone | 2 | 3
  Tramadol | 2 | 3
  Oxycodone hydrochloride | 1 | 2
  Codeine | 1 | 0
  Hydromorphone hydrochloride | 0 | 1
  Tramadol hydrochloride | 0 | 1

23. Secondary Outcome: Number of Participants With Abnormal Laboratory Blood Chemistry Values
Description: Participants with abnormal chemistry values as assessed by the investigator are reported here. The marked reference range are as follows: calcium <1.12 or > 1.47 millimoles per liter (mmol/L) and sodium < 130 or > 150 mmol/L.
Time Frame: At Screening and Day 3
Population: Safety population consisted of all participants who received at least 1 dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 20
Participants
  Screening: Calcium, Ionized (mmol/L): High > 1.47 | 1 | 0
  Day 3: Calcium, Ionized (mmol/L): Low < 1.12 | 0 | 1
  Day 3: Sodium (mmol/L): Low < 130 | 0 | 1

24. Secondary Outcome: Number of Participants With Abnormal Laboratory Hematology Values
Description: Participants with abnormal hematology values as assessed by the investigator are reported here. Hematology abnormalities were only observed on Day 3. The marked reference range are as follows: hematocrit < 30 or > 58%, hemoglobin < 10 or > 20 grams per deciliter (g/dL) and Lymphocytes/Leukocytes < 10 or > 60%.
Time Frame: Day 3
Population: Safety population consisted of all participants who received at least 1 dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 20
Participants
  Day 3: Hematocrit (%): Low < 30 | 6 | 1
  Day 3: Hemoglobin (g/dL): Low < 10 | 8 | 4
  Day 3: Lymphocytes/Leukocytes (%): Low < 10 | 3 | 3

25. Secondary Outcome: Number of Participants With Abnormal Laboratory Coagulation Values
Description: Participants with abnormal coagulation values as assessed by the investigator are reported here. The marked reference range are as follows: prothrombin international normalized ratio > 1.3, prothrombin time > 20 seconds, and activated partial thromboplastin time > 45 seconds.
Time Frame: At Screening and Day 3
Population: Safety population consisted of all participants who received at least 1 dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 20
Participants
  At Screening: Prothrombin International Normalized Ratio: High > 1.3 | 1 | 1
  At Screening: Prothrombin Time (seconds): High > 20 | 1 | 0
  Day 3: Activated Partial Thromboplastin Time (seconds): High > 45 | 0 | 2
  Day 3: Prothrombin International Normalized Ratio: High > 1.3 | 4 | 3
  Day 3: Prothrombin Time (seconds): High > 20 | 2 | 3

26. Secondary Outcome: Number of Participants With Abnormal Laboratory Urinalysis Values
Description: Participants with abnormal urinalysis values as assessed by the investigator are reported here. The normalized estimated glomerular filtration rate (eGFR) values were (mL/min/surface area (SA)) < 55.
Time Frame: At Screening and Day 3
Population: Safety population consisted of all participants who received at least 1 dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 20
Participants | 0 | 0

27. Secondary Outcome: Number of Participants With Abnormal Vital Signs: Blood Pressure Measurements
Description: Participants with abnormal blood pressure measurements as assessed by the investigator are reported here. The following parameters were considered in the assessment of abnormal blood pressure measurements: systolic blood pressure >180 millimeters of mercury (mmHg); systolic blood pressure > 200 mmHg; diastolic blood pressure < 50 mmHg.
Time Frame: Pre-infusion at Days 1, 2 (Pre and Postoperative) and 3; At Post infusion on Day 1 (15, 30, 45, 60 mins); Day 2 Preoperative (15, 30, 45 mins); Postoperative (30 mins); Day 3 (15 and 30 mins); and 30 mins after end of each infusion
Population: Safety population included all participants who received at least 1 dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 20
Participants
  Systolic Blood Pressure > 180 mmHg: On Day 1 (Prior to Infusion) | 1 | 1
  Systolic Blood Pressure > 180 mmHg: On Day 1 (30 Minutes After End of Infusion) | 1 | 0
  Systolic Blood Pressure > 180 mmHg: On Day 2 Preoperative (Prior to Infusion) | 1 | 1
  Systolic Blood Pressure > 180 mmHg: On Day 2 Preoperative (15 Minutes Post Infusion) | 1 | 1
  Systolic Blood Pressure > 180 mmHg: On Day 2 Preoperative (30 Minutes Post Infusion) | 1 | 2
  Systolic Blood Pressure > 180 mmHg: On Day 2 Preoperative (45 Minutes Post Infusion) | 2 | 1
  Systolic Blood Pressure > 180 mmHg: On Day 2 Postoperative (Prior to Infusion) | 1 | 0
  Systolic Blood Pressure > 200 mmHg: On Day 2 Preoperative (15 Minutes Post Infusion) | 0 | 1
  Systolic Blood Pressure > 200 mmHg: On Day 2 Preoperative (30 Minutes Post Infusion) | 0 | 1
  Diastolic Blood Pressure < 50 mmHg: On Day 1 (Prior to Infusion) | 0 | 1
  Diastolic Blood Pressure < 50 mmHg: On Day 1 (15 Minutes Post Infusion) | 0 | 1
  Diastolic Blood Pressure < 50 mmHg: On Day 1 (30 Minutes Post Infusion) | 0 | 1
  Diastolic Blood Pressure < 50 mmHg: On Day 1 (45 Minutes Post Infusion) | 1 | 0
  Diastolic Blood Pressure < 50 mmHg: On Day 1 (60 Minutes Post Infusion) | 1 | 0
  Diastolic Blood Pressure < 50 mmHg: On Day 1 (30 Minutes After End of Infusion) | 0 | 1
  Diastolic Blood Pressure < 50 mmHg: On Day 2 Preoperative (30 Minutes After End of Infusion) | 1 | 2
  Diastolic Blood Pressure < 50 mmHg: On Day 2 Postoperative (30 Minutes Post Infusion) | 0 | 1
  Diastolic Blood Pressure < 50 mmHg: On Day 3 (Prior to Infusion) | 1 | 0
  Diastolic Blood Pressure < 50 mmHg: On Day 3 (15 Minutes Post Infusion) | 0 | 1
  Diastolic Blood Pressure < 50 mmHg: On Day 3 (30 Minutes Post Infusion) | 1 | 0
  Diastolic Blood Pressure < 50 mmHg: On Day 3 (30 Minutes After End of Infusion) | 1 | 0

28. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameter: Heart Rate
Description: A 12-lead ECG was to be performed to obtain heart rate. The baseline was defined as Day 1 pre-infusion measurement.
Time Frame: Baseline (Day 1 pre-infusion); Day 3 pre and post-infusion
Population: Safety population included all participants who received at least 1 dose of the study treatment. Number analyzed is the number of participants available for analysis at the specified time points.
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 20
beats/minute
  At Baseline | 63.7 (7.05) | 64.5 (11.24)
  Change From Baseline on Day 3 (Prior to Infusion): number analyzed (Participants) | 18 | 19
  Change From Baseline on Day 3 (Prior to Infusion) | 1.2 (9.16) | 5.1 (11.08)
  Change From Baseline on Day 3 (Post Infusion): number analyzed (Participants) | 17 | 19
  Change From Baseline on Day 3 (Post Infusion) | 8.4 (7.73) | 5.7 (11.96)

29. Secondary Outcome: Change From Baseline in ECG Parameters: QT Interval and QT Interval Corrected by the Fridericia Formula (QTcF)
Description: A 12-lead ECG was performed after the participant had rested quietly for at least 5 minutes in a supine or sitting position. The parameters evaluated from the participant ECG trace included QT interval and QTc (corrected). Corrected QTc intervals were calculated using Fridericia's correction formula. The baseline was defined as Day 1 pre-infusion measurement.
Time Frame: Baseline (Day 1 pre-infusion); Day 3 pre and post-infusion
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 20
msec
  QT Interval: At Baseline | 422.1 (31.13) | 408.9 (26.02)
  QT Interval: Change From Baseline on Day 3 (Prior to Infusion): number analyzed (Participants) | 18 | 19
  QT Interval: Change From Baseline on Day 3 (Prior to Infusion) | 2.6 (36.64) | -9.3 (37.04)
  QT Interval: Change From Baseline on Day 3 (Post Infusion): number analyzed (Participants) | 17 | 19
  QT Interval: Change From Baseline on Day 3 (Post Infusion) | -24.3 (22.52) | -15.6 (31.01)
  QTcF: At Baseline | 429.1 (22.38) | 416.4 (16.68)
  QTcF: Change From Baseline on Day 3 (Prior to Infusion): number analyzed (Participants) | 18 | 19
  QTcF: Change From Baseline on Day 3 (Prior to Infusion) | 6.4 (22.48) | -1.3 (23.71)
  QTcF: Change From Baseline on Day 3 (Post Infusion): number analyzed (Participants) | 17 | 19
  QTcF: Change From Baseline on Day 3 (Post Infusion) | -7.3 (15.08) | -4.1 (14.91)

30. Primary Outcome: Effect of GRF6021 on Immune Responses to Surgery as Determined by Cytometry by Time of Flight (CyTOF) on Day 3
Description: as for outcome 1
Time Frame: Day 3
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: predicted value
Arm/Group | GRF6021 | Placebo
Number analyzed (Participants) | 18 | 18
predicted value | 0.7829 [0.5941 to 0.8824] | 0.2871 [0.1201 to 0.7090]

ADVERSE EVENTS:
Time Frame: From Baseline (Day -7 to -3 prior to surgery) up to end of study (approximately Day 46)
Description: Safety population included all participants who received at least 1 dose of the study treatment.
Groups:
- GRF6021: Participants received 4 doses of GRF6021, 250 mL, IV infusion. The first dose was administered on day before surgery, the next two doses on the day of surgery i.e., within 4 hours before start of surgery (first incision), and then upon arrival in the postoperative care unit (within 5 hours after the first incision) and the finally last dose was administered on the day after the surgery.
Arm/Group | GRF6021 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/20
Other Adverse Events (participants affected / at risk) | 14/18 | 14/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GRF6021 (N=18) | Placebo (N=20)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Eye irritation (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 7 | 5
Chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Stitch abscess (Infections and infestations) | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Incision site erythema (Injury, poisoning and procedural complications) | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 3 | 0
Blood pressure increased (Investigations) | 0 | 1
Gamma-glutamyl transferase increased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement contains language that restricts the PI from discussing or publishing Sponsor confidential and/or proprietary information. The embargo period may be extended by mutual agreement of the Sponsor and PI.

DOCUMENTS (3):
  • Study Protocol (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT03981419/Prot_000.pdf
  • Statistical Analysis Plan: Original Statistical Analysis Plan (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT03981419/SAP_001.pdf
  • Statistical Analysis Plan: Supplementary Statistical Analysis Plan (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT03981419/SAP_002.pdf